CLINICAL TRIAL: NCT04926441
Title: Stress Levels and Mental Well-Being Among Polish, Slovakian and Lithuanian Students During E-learning
Brief Title: Stress Levels and Mental Well-Being Among Students During e-Learning
Status: Completed | Type: Observational
Sponsor: The Opole University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: COVID_International
Record Dates: First submitted 2021-06-13; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Anxiety; Depression
Keywords: depression; anxiety; COVID-19; e-Learning
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students from 8 European Universities, regardless of field of study and academic year: At the beginning of the summer semester of the 2020/2021 academic year, stress levels as well as symptoms of anxiety and depression were assessed in students at four universities.
  Interventions: Diagnostic Test: Stress Levels and Mental Well-Being assessment

INTERVENTIONS:
Diagnostic Test: Stress Levels and Mental Well-Being assessment — At the beginning of the summer semester of the 2020/2021 academic year, stress levels as well as symptoms of anxiety and depression were assessed in students at four universities.

SUMMARY:
Introducing restrictions on human contact has been effective in preventing the uncontrolled spread of COVID-19, however, it appears to have negatively impacted mental health. Psychological problems in different age groups occur with different intensity and duration of the pandemic. This study was aimed to assess the impact of introducing distance learning (e-Learning) on the stress levels and mental well-being among Polish, Slovak and Lithuanian Students.

DETAILED DESCRIPTION:
The COVID-19 pandemic has had the effect of accelerating changes in educational processes around the world. It resulted in a rapid conversion from face-to-face to online classes. This has disrupted the regular pattern of education and standard practices that have been followed for many years. It is a big organizational challenge for the academics but most importantly for the students. Remote learning has resulted in long-term social isolation and limitations in interaction with peers. It has also been noted that about 30% of students have symptoms of depression and increased levels of perceived stress, which during the COVID-19 pandemic affects about 50% of young people. Many factors have an impact on this condition, besides the epidemic situation, the social mood and the numerous restrictions, the prolonged time spent online and the reduced level of physical activity have an additional negative impact on their mental health. Due to the dynamic situation of the pandemic, there is a lack of current studies on the mental state of young people especially in the context of ongoing e-learning. Therefore, it was decided to investigate what is the prevalence of depressive disorders and the level of perceived stress during the ongoing remote learning in the group of students of 8 European Universities among Poland, Slovakia and Lithuania.

ELIGIBILITY:
Inclusion Criteria:

* Students attending the course cycle

Exclusion Criteria:

* Inability to self-complete the research questionnaires;
* Psychiatric or psychological treatment, likewise taking medications that affect the psyche during the research project;

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students participating in active learning
Sampling Method: Probability Sample
Enrollment: 4870 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Perception of Stress Questionnaire (PSQ) | 20 minutes
  The Perception of Stress Questionnaire (PSQ) is a 27-item scale scoring from 1 to 5 for each item. 21 items examine the level of stress in the area of emotional tension, external stress and intrapsychic stress, and 6 items refer to the lie scale. The global scoring for perception of stress ranges from 21 to 105 with a cut-off point of 60 for high level of perceived stress. The higher the score, the greater the sense of stress. PSQ will be performed at the beginning and after four weeks of treatment.
Beck's Depression Inventory | 20 minutes
  The BDI-II is a tool used to determine the degree of intensity of depressive symp-toms. The 21-item questionnaire consists of two parts: emotional and somatic. Depending on the number of points obtained, the severity of depression can be assessed. A range of 0-10 points indicates no depression, 11-27 indicates moderate mood disorder, and 28 indicates major depressive disorder. The cutoff for dividing patients into depressive and non-depressive subgroups was a score of 10, following the guidelines given by Beck et al.
Authors' survey | 10 minutes
  The survey contains five sections on the impact of e-learning on various aspects of life. The survey responses were structured on a 5-point Likert scale from 1 to 5, where 1 refers to "strongly disagree" statement and 5 to "definitely agree". Questions were grouped into areas: Social life (3 questions), Education skills (4 questions), Eco-nomic field (2 questions), Nutrition habits and drugs (2 questions). The questionnaire showed satisfactory reliability with a Cronbach alpha of 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Szczepańska-Gieracha, Prof, Study Director — The University School of Physical Education in Wroclaw; Anna Rutkowska, PhD, Principal Investigator — The Opole University of Technology
Locations (8):
- Lithuanian Sports University, Kaunas, Lithuania
- Poland (3):
  - Jan Dlugosz University in Czestochowa, Częstochowa
  - Faculty of Physical Education and Physiotherapy, Opole University of Technology, Opole
  - The University School of Physical Education in Wroclaw, Wroclaw
- Slovakia (4):
  - Slovak Medical University in Bratislava, Banská Bystrica
  - Matej Bel University, Banská Bystrica
  - Technical University of Košice, Košice
  - Constantine the Philosopher University in Nitra, Nitra

IPD SHARING:
Plan to Share IPD: No